CLINICAL TRIAL: NCT02896231
Title: A Phase I Open-label, Multicenter Dose Escalation Study to Assess the Safety, Tolerability and Pharmacokinetics (PK) of PLB1001 in Patients With Met-positive (Met+) Advanced Non-small Cell Lung Cancer (NSCLC)
Brief Title: First-in-human Phase I Study of a Selective c-Met Inhibitor PLB1001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Pearl Biotechnology Limited Liability Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMO-PLB1001-2013012-01
Record Dates: First submitted 2016-08-16; First posted 2016-09-12 (Estimated); Last update posted 2019-11-22 (Actual); Status verified 2017-10

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PLB1001 (Experimental): There are 5 dose cohorts, including 50mg BID, 100mg BID, 150mg BID, 200mg BID and 275mg BID in the dose escalation stage and PLB1001 will be administered orally to patients twice daily for each dose cohort.
  Interventions: Drug: PLB1001

INTERVENTIONS:
Drug: PLB1001 — PLB1001 is a capsule in the form of 25 mg and 100mg, twice daily.
  Other Names: Bozitinib

SUMMARY:
This phase I, first-in-human dose-escalation study was conducted to determine the maximum tolerated dose (MTD), recommended phase II dose (RP2D), dose-limiting toxicities (DLTs), pharmacokinetics (PK) profile, and preliminary antitumor activity of PLB1001.

DETAILED DESCRIPTION:
This is a Phase I, open-label, multicentre study of PB1001 administered orally to patients with Met-positive (Met+) advanced NSCLC. The study includes a Dose-escalation Part (part A)and a Dose Expansion Part(part B). The aim of the part A is to estimate the MTD and to identify the dose limited toxicity(DLT) and the recommended phase II dose (RP2D) for PLB1001 single agent as well as to determine the PK/PD profile .Once response has been observed in certain dose level ,then followed by the expansion part to further assess the clinical efficacy and safety of PLB1001 single agent. Aprox. 40 patients will be enrolled in PART A, while 20-30 patients for expansion cohort .

PLB1001 is a potent selective c-Met inhibitor. PLB1001 acts on cancer by blocking abnormal cmet-mediated signalling, leading to profound tumour growth inhibition in xenografts of non-small cell lung cancer (NSCLC) tumours. Preliminary data from a c-Met inhibitor INC 280 has provided possibility on the safety and clinical activity of PLB1001 monotherapy in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Age≥18 years
* Histologically or cytologically confirmed advanced non-small cell lung cancer
* Must have evidence of c-Met positivity from the results of molecular pre-screening evaluations
* At least one measurable lesion as per RECIST v1.1
* Patients must have recovered from all toxicities related to prior anticancer therapies to grade ≤ 1
* ECOG Performance Status of 0-2

Exclusion Criteria:

* Previous or current treatment with a c-Met inhibitor or HGF-targeting therapy
* Symptomatic central nervous system (CNS) metastases that are neurologically unstable or requiring increasing doses of steroids to control, and patients with any CNS deficits.
* Clinically significant, uncontrolled heart diseases. Unstable angina History of documented congestive heart failure (New York Heart Association functional classification > II) Uncontrolled hypertension defined by a Systolic Blood Pressure (SBP) ≥ 140 mm Hg and/or Diastolic Blood Pressure (DBP) ≥ 90 mm Hg Arrhythmias
* Active peptic ulcer disease or gastritis
* Adverse events from prior anti-cancer therapy that have not resolved to Grade ≤ 1, except for alopecia
* Major surgery within 4 weeks prior to starting PLB1001
* Previous anti-cancer and investigational agents within 4 weeks before first dose of PLB1001. If previous treatment is a monoclonal antibody, then the treatment must be discontinued at least 6 weeks before first dose of PLB1001.
* Pregnant or nursing women
* Involved in other clinical trials < 30 days prior to Day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-04; Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with dose-limiting toxicities | 2 years

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of PLB1001 and its metabolite | Day 1-2 Single Dose and Day 1-28 Steady State
  In the study of single-dose, full Pharmacokinetics (PK) profiles ofPLB1001 will be obtained following administration of a single oral dose of PLB-1001 on Day 1 to Day 2. At multiple-dose, Pharmacokinetics (PK) sampling will include a pre-dose and at the 0.5, 2, 4, 6, 8, 10, 10.5, 12 and 13 hour time points on days 8, 22of dosing in the first 28-Day cycle of therapy, and pre-dose on days 9, 14, 15, 16and 23 of the first 28-Day cycle of therapy
Maximum plasma concentration observed (Cmax) of PLB1001 and its metabolite | Day 1-2 Single Dose and Day 1-28 Steady State
  In the study of single-dose, full Pharmacokinetics (PK) profiles ofPLB1001 will be obtained following administration of a single oral dose of PLB-1001 on Day 1 to Day 2. At multiple-dose, Pharmacokinetics (PK) sampling will include a pre-dose and at the 0.5, 2, 4, 6, 8, 10, 10.5, 12 and 13 hour time points on days 8, 22of dosing in the first 28-Day cycle of therapy, and pre-dose on days 9, 14, 15, 16and 23 of the first 28-Day cycle of therapy
Time to Cmax (Tmax) of PLB1001 and its metabolite | Day 1-2 Single Dose and Day 1-28 Steady State
  In the study of single-dose, full Pharmacokinetics (PK) profiles ofPLB1001 will be obtained following administration of a single oral dose of PLB-1001 on Day 1 to Day 2. At multiple-dose, Pharmacokinetics (PK) sampling will include a pre-dose and at the 0.5, 2, 4, 6, 8, 10, 10.5, 12 and 13 hour time points on days 8, 22of dosing in the first 28-Day cycle of therapy, and pre-dose on days 9, 14, 15, 16and 23 of the first 28-Day cycle of therapy
Preliminary antitumor activity of PLB1001 | 2 years
  Preliminary antitumor activity of PLB1001 assessed using RECIST1.1

CONTACTS AND LOCATIONS:
Overall Officials: Yilong Wu, MD, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided